CLINICAL TRIAL: NCT05531487
Title: MC-career Choice Questionnaire for Exploring Insights Regarding the Motivations of Chinese Medical Students.
Brief Title: A 14-item Questionnaire Regarding Career Preferences Among Chinese Medical Undergraduate Students.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, YIZHUO GAO, Doctor, Shengjing Hospital
Other Study IDs: MC-career choice
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Career Burnout; Student Burnout
Keywords: career choice; medical students
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical students: Undergraduate medical students at one Medical University.
  Interventions: Other: Questionnaire Survey

INTERVENTIONS:
Other: Questionnaire Survey — All students received a 'QR code' link to the survey.

SUMMARY:
This survey was performed as part of a career choice research program for undergraduate medical students. All students received a QR code link to the survey as part of their course work.

DETAILED DESCRIPTION:
This survey was performed as part of a career choice research program for undergraduate medical students. All students received a QR code link to the survey as part of their course work, although participation was voluntary and anonymous. All participants received verbal and online explanations of the questionnaire and were informed that informed consent would be assumed if they completed and submitted the questionnaire. The questionnaire was administered, and data were collected using a free online tool.

ELIGIBILITY:
Inclusion Criteria:

* Participants from several four-year student classes medical students were enrolled.

Exclusion Criteria:

* Students who did not complete or declined to complete the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cross-sectional survey was supposed to be conducted. Participants from eight fourth-year student classes who were studying clinical medicine were enrolled.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire Results | 14 days
  The questionnaire was administered, and data were collected using a free online tool.This score was a 7 point likert scale questionnaire, the minimum value was 1 and maximum value was 7, higher scores mean a stronger attitude.

CONTACTS AND LOCATIONS:
Overall Officials: DONG JIA, Principal Investigator — Shengjing Hospital
Locations (1):
- Shenjing Hospital of CHINA MEDICAL UNIVERSITY, Shenyang, Liaoning, China